CLINICAL TRIAL: NCT05641883
Title: A Prospective Pilot Study of the Combination of CardiaMend and Amiodarone for the Prevention of Postoperative Atrial Fibrillation (POAF) in Patients Undergoing Isolated Coronary Artery Bypass Grafting or Isolated Valve Surgery
Brief Title: CardiaMend and Amiodarone for the Prevention of POAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saint Alphonsus Regional Medical Center (Other)
Responsible Party: Principal Investigator, Robert Saeid Farivar, MD, Medical Director of Cardiothoracic Surgery, Saint Alphonsus Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00066172
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: POAF; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): All eligible patients that are enrolled with receive the CardiaMend patch soaked in amiodarone
  Interventions: Combination Product: CardiaMend with antiarrhythmic

INTERVENTIONS:
Combination Product: CardiaMend with antiarrhythmic — Pericardial patch with antiarrhythmic drug (amiodarone) topically applied

SUMMARY:
The principal purpose of this investigator-initiated trial is to study the use of the CardiaMend device soaked in the anti-arrhythmic drug amiodarone, and how it may decrease the development of atrial fibrillation in patients that have undergone a coronary artery bypass surgery, or isolated valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-85 years
* Able to provide written informed consent, understand and be willing to comply with study-related procedures.
* Scheduled to undergo open-chest cardiac surgery via complete median sternotomy for coronary artery bypass graft (CABG), or isolated valve repair/replacement.
* Inclusionary valve repair/replacement procedures with the primary reason for surgery inclusive of aortic valve repair/replacement or mitral valve repair/replacement.
* Left atrial appendage (LAA) procedures are allowed if CABG and/or valve repair or replacement is the qualifying surgical procedure, but is not a qualifying surgical procedure on its own.
* In sinus rhythm at the time of consultation and on a previous EKG, or no history of atrial fibrillation (note: continuous ECG monitoring for 48 hours is not required)

Exclusion Criteria:

* Unable to give voluntary written informed consent, is unlikely to cooperate or is legally incompetent, including subjects who are institutionalized by court or official order, or in a dependency relationship with testing center or investigator.
* Any condition which could interfere with the subject's ability to comply with the study.
* Ongoing participation in an interventional clinical study or during the preceding 30 days.
* Female subjects who are pregnant, breastfeeding, were pregnant within the last three months or are planning a pregnancy during the course of the study.
* Active skin or deep infection at the site of implantation.
* History of chronic wounds or wound-healing disorders.
* Known connective tissue diseases (e.g. Ehlers-Danlos syndrome, Epidermolysis bullosa, Marfan syndrome, Osteogenesis imperfecta).
* Immune-suppressed subjects, immune-deficiency subjects (properly managed diabetes mellitus is not an exclusion criterion).
* The subject has an implantable cardiac device (i.e., cardiac resynchronization therapy devices with and without defibrillator capabilities (CRTs and CRT-Ds), implantable cardioverter-defibrillators (ICD) and pacemakers).
* Known history of atrial fibrillation (in any form including paroxysmal atrial fibrillation).
* History of ablation for atrial fibrillation.
* Patients already receiving amiodarone as a treatment for atrial fibrillation or ventricular arrhythmias during the procedure.
* Disease of the left pleura, previous intervention in the left pleural space, or chest deformity.
* Subjects with end-stage chronic-renal disease / dialysis.
* Subjects with heart failure (BNP>1000), low ejection fraction (<35%), end stage renal disease (on dialysis or creatinine >1.8).
* STS risk >5.5% for 30 day mortality.
* Patients electing to receive an ablative procedure for atrial fibrillation.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of POAF | 5 days
  Incidence of POAF up to patient discharge as defined as atrial fibrillation/flutter (AF) after OR exit that lasted longer than one hour, or lasted less than one hour but required medical or procedural intervention.

SECONDARY OUTCOMES:
Time until discharge | 5 days
  Burden of atrial fibrillation as defined by additional treatment regimen, additional time in ICU, and/or complications directly associated with atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Saeid Farivar, MD, PhD, Principal Investigator — Saint Alphonsus Regional Medical Center

IPD SHARING:
Plan to Share IPD: No